CLINICAL TRIAL: NCT01261780
Title: Treatment of Painful Chemotherapy -Induced Peripheral Neuropathy With the MC-5A Pain Therapy Medical Device, a Randomized, Double-Blind, Sham-Controlled Clinical Trial
Brief Title: MC-5A for Chemotherapy Induced Peripheral Neuropathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: OS10328; 2010-0361 (Other: Institutional Review Board); NCI-2012-00075 (Registry Identifier: NCI Trial ID); A534260 (Other: UW Madison); SMPH\MEDICINE\HEM-ONC (Other: UW Madison)
Record Dates: First submitted 2010-12-09; First posted 2010-12-16 (Estimated); Results first posted 2017-11-06 (Actual); Last update posted 2019-12-02 (Actual); Status verified 2017-10

CONDITIONS: Neuropathy, Paraneoplastic
Keywords: neuropathy,paraneoplastic; paraneoplastic peripheral neuropathy; pain; hyperalgesia
MeSH Terms: conditions — Paraneoplastic Polyneuropathy; Pain; Hyperalgesia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sham device (Sham Comparator): Sham therapy device to area of painful chemotherapy induced peripheral neuropathy (CIPN) for 45 minutes daily x 10 days
  Interventions: Drug: Sham device
- MC-5A treatment (Active Comparator): MC-5A therapy to the area of painful CIPN for 45 minutes daily for a total of 10 days.
  Interventions: Device: MC-5A

INTERVENTIONS:
Device: MC-5A — 45 minutes daily x 10 treatments (given over the course of 2 weeks)
  Other Names: Scrambler therapy
  Arms: MC-5A treatment
Drug: Sham device — Sham therapy daily x 45 minutes for 10 treatments (given over course of 2 weeks)
  Other Names: TRA-1
  Arms: Sham device

SUMMARY:
Painful chemotherapy induced peripheral neuropathy (CIPN) is a common complication of cancer therapy with few treatment options. CIPN is a complex side effect that varies between individuals and can be difficult to describe, difficult to treat and can significantly effect quality of life for patients.

The purpose of this study is to determine if patients with painful CIPN will have a decrease in pain scores after treatment with the MC-5A device.

ELIGIBILITY:
Inclusion Criteria:

* painful peripheral neuropathy resulting from chemotherapy
* pain must be present for minimum of 6 months
* must be able to read/understand English
* stable analgesics regimens allowed (no change for past 7 days)

Exclusion Criteria:

* painful peripheral neuropathy that is not the result of chemotherapy
* pregnant women
* patients unable to wean off anti-epileptics
* patients currently receiving chemotherapy known to cause peripheral neuropathy
* patients with pacemakers or implanted defibrillators
* patients with vena cava or aneurysm clips
* patients with a history of epilepsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2011-04; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tony Campbell, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin, United States

REFERENCES:
- See also: University of Wisconsin Carbone Cancer Center — https://cancer.wisc.edu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study enrolled patients from May 2011 through May 2012 at a large research university.
Period: Overall Study
Arm/Group | Sham Device | MC-5A Treatment
Started | 7 | 7
Completed | 5 | 5
Not Completed | 2 | 2
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Event not related to subject | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sham Device | MC-5A Treatment | Total
Number analyzed (Participants) | 7 | 7 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 3 | 9
  >=65 years | 1 | 4 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 8
  Male | 2 | 4 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 7 | 7 | 14
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 7 | 7 | 14
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 7 | 14

OUTCOME MEASURES:

1. Primary Outcome: Change in Mechanical Visual Analog Scale (mVAS) Using Quantitative Sensory Pain Testing (QSPT)
Description: Pain levels will be compared as measured by changes in mVAS, and quantified and tested for normal distribution. If normally distributed, parametric test (i.e., two-sample t-test) will be used; p-values <0.05 will be considered statistically significant. If changes in mVAS are not normally distributed, non-parametric testing such as Wilcoxon rank-sum will be performed. VAS is measured at 3 time points.
  mVAS and deficits scale are used to obtain continuous quantitative information about positive and negative sensory phenomena during application of QSPT stimulation.
  Patients provide rating of positive sensory phenomena using mVAS if the stimulus at the pain test site is increased or painful when compared to normal control site. Rating on mVAS is obtained by instructing the patient to pull out the mechanical scale with millimeters (looks like a slide ruler) to reflect intensity of any painful sensation on a scale of 0 - 10, with 10 being the worst. Score = Visit - Baseline.
Time Frame: Baseline, Visit 1 (Day 1), Vist 10 (Day 10), and End of Study (Week 12, +/- 2 weeks)
Population: The number analyzed differs per row as some participants dropped out or did not receive all 10 treatments. For example, on the Sham Device arm, only 4 participants were treated on day 10 but 5 returned for the final visit. Because this was a pilot study, all participant data was analyzed and is included here.
Measure: Mean (Standard Deviation); unit: Millimeters
Arm/Group | Sham Device | MC-5A Treatment
Number analyzed (Participants) | 7 | 6
Millimeters
  Visit 1 (Day 1) | 5.14 (29.1) | -2.00 (17.0)
  Visit 10 (Day 10): number analyzed (Participants) | 4 | 5
  Visit 10 (Day 10) | 1.25 (2.50) | 6.76 (24.7)
  End of Study (Week 12, +/- 2 weeks): number analyzed (Participants) | 5 | 6
  End of Study (Week 12, +/- 2 weeks) | -11.2 (5.36) | 3.80 (3.42)

2. Secondary Outcome: Adverse Events
Description: The number of participants experiencing adverse events, as defined by CTCAE
Time Frame: Up to 3 months
Measure: Number; unit: participants
Arm/Group | Sham Device | MC-5A Treatment
Number analyzed (Participants) | 7 | 7
participants | 4 | 4

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for up to 3 months.
Description: This study uses the CTCAE v.4 definition of adverse event, which does not differ from the clinicaltrials.gov definitions.
Arm/Group | Sham Device | MC-5A Treatment
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/7
Serious Adverse Events (participants affected / at risk) | 1/7 | 0/7
Other Adverse Events (participants affected / at risk) | 4/7 | 4/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sham Device (N=7) | MC-5A Treatment (N=7)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sham Device (N=7) | MC-5A Treatment (N=7)
Anxiety (Psychiatric disorders) | 0 | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0
Fatigue (General disorders) | 0 | 1 (2)
Gait disturbance (General disorders) | 0 | 1 (1)
Hypertension (Vascular disorders) | 3 (3) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 | 1 (1)
Pain (General disorders) | 1 (1) | 2 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0
Skin, Other - Scratch in area by knee (Skin and subcutaneous tissue disorders) | 1 (1) | 0
Skin, Other - Basel Cell Cancer Removed (Skin and subcutaneous tissue disorders) | 0 | 1 (1)
Skin, Other - Redness at site of electrode pads (1 hr post treatment) (Skin and subcutaneous tissue disorders) | 1 (1) | 0

LIMITATIONS AND CAVEATS:
The small sample size is subject to type II error. The estimated effect size for MC5A is high: the company estimates 100% of patients will respond. Thus our power calculations suggested a small sample could still detect a difference.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes